CLINICAL TRIAL: NCT00454025
Title: Intraocular Pressure Changes Associated With Muslim Prayer Postural Changes
Brief Title: Intraocular Pressure (IOP) Changes Associated With Muslim Prayer Postural Changes
Status: Terminated | Type: Observational
Why Stopped: Stopped due to low enrollment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 06-1015
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Glaucoma
Keywords: glaucoma; intraocular pressure; postural changes
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma: Patients with Glaucoma
- Healthy Patients: Patients without glaucoma

SUMMARY:
Elevated intraocular pressure is widely accepted as a risk factor for glaucoma and controlling the pressure remains the cornerstone of effective treatment. There is evidence that posture can have a significant effect on intraocular pressure fluctuations. Salat (or Salah) refers to the five daily prayers performed by Muslims. The time spent praying in a kneeling or prostrate position may be associated with wide fluctuations in intraocular pressure, potentially sight-threatening for Muslim patients with glaucoma. The researchers seek to investigate the link between traditional daily Muslim prayer postural changes and intraocular pressure changes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open angle glaucoma
* Must be age 18 and up
* Provide written informed consent to participate
* Able to cooperate with ocular examination for 60-90 minutes
* Able to assume the standing, bowing, and prostrate positions

Exclusion Criteria:

* Special patient populations (children, pregnant women, prisoners etc.)
* Patients who have had glaucoma surgery that could effect the change in intraocular pressure (ie trabeculectomy, tube-shunts, etc.)
* Patients who are unable to assume bowing or kneeling positions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 and up, diagnosed with primary open angle glaucoma, and are able to assume the standing, bowing, and prostrate positions.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | Single Exam

SECONDARY OUTCOMES:
Positional Intraocular Pressure Changes | Single Exam

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — Rocky Mountain Lions Eye Institute
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States